CLINICAL TRIAL: NCT05154383
Title: Effect of High-Dose Quadrivalent Influenza Vaccine (Efluelda®) Versus Standard-Dose (QIV-SD), in Subjects 65 Years of Age and Older on Innate Immunity, Including Gene Expression
Acronym: INFLUOMICS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Euraxi Pharma (Industry); Hospices Civils de Lyon (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-05
Record Dates: First submitted 2021-11-03; First posted 2021-12-13 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2021-11

CONDITIONS: Vaccine Reaction
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose Quadrivalent Influenza Vaccine (Experimental): One injection of the high-dose Efluelda vaccine will be given to the patient
  Interventions: Biological: Experimental arm : High-Dose Quadrivalent Influenza Vaccine (Efluelda)
- Standard-Dose Quadrivalent Influenza Vaccine (Active Comparator): One injection of the standard-dose Influvactetra vaccine will be given to the patient
  Interventions: Biological: Active Comparator: Standard-Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Experimental arm : High-Dose Quadrivalent Influenza Vaccine (Efluelda) — Patient will received one dose of High Dose Quadrivalent Influenza Vaccine according to marketing authorization.
  Arms: High-Dose Quadrivalent Influenza Vaccine
Biological: Active Comparator: Standard-Dose Quadrivalent Influenza Vaccine — Patient will received one dose of Standard Dose Quadrivalent Influenza Vaccine according to marketing authorization.
  Arms: Standard-Dose Quadrivalent Influenza Vaccine

SUMMARY:
The purpose of the study is to evaluate innate and adaptive immunity following QIV-HD vaccination compared to QIV-SD vaccination in people 65 years of age and older.

DETAILED DESCRIPTION:
The hypothesis is that higher dose of antigen can increase the intensity and the quality of innate immunity, as the adaptive humoral and cellular responses.

In this study, the objectif is to evaluate innate and adaptive immunity following QIV-HD vaccination compared to QIV-SD vaccination in people 65 years of age and older.

Modifications of early blood molecular (transcriptome) and cellular (blood phenotyping) signatures within the first 24 hours following vaccination will be investigated. The association between early gene signature and late influenza-specific humoral immune responses weeks/months after vaccination will be also assessed.

This study is a hase IV, randomized, open-label, active-controlled, multi-center study comparing the immune response induced by QIV-HD vaccine (intervention) and QIV-SD vaccine (control).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 years or older, the day of inclusion;
2. Have signed and dated Informed Consent Form;
3. Able and willing to attend all scheduled visits, and to comply with study procedures;
4. Covered by French health insurance.

Non-Inclusion Criteria :

1. Any vaccine injection (including COVID-19 vaccine) in the 4 weeks preceding study inclusion;
2. Plan to receive any vaccine (including COVID-19 vaccine) in the 4 weeks following study inclusion;
3. Already vaccinated against influenza for 2021-2022 season;
4. Hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances;
5. HIV infection;
6. Active Hepatitis B, or active Hepatitis C;
7. Previous Guillain Barré syndrome;
8. Ongoing immunosuppressive treatment or active immunodeficiency;
9. Receipt of immune globulins, blood or blood-derived products in the past 3 months;
10. Thrombocytopenia or bleeding disorder, receipt of anticoagulants contraindicating IM vaccination based on investigator's judgment;
11. Influenza-like illness symptoms, including COVID-19, within 4 weeks before study inclusion;
12. Personnes referred to in articles L1121-6 and L1121-8 of Public Health Code (persons deprived of liberty by judicial or administrative decision and persons subject to a legal protection measure: guardianship or curatorship).

Exclusion Criteria:

1. Any subject presenting with influenza-like illness symptoms, including COVID-19 between inclusion (visit 1) and randomization (visit 2);
2. Subject unable to attempt visit at Day 0 (visit 2) and Day 1 (visit 3);
3. Blood sample at Day 0 (visit 2) impossible to obtain;
4. Receipt of vaccine injection or equivalent between inclusion (visit 1) and randomization (visit 2), other than those allowed and planned in the study. This includes non-study dose of 2021-2022 influenza vaccine, blood-derived immune globulins, blood, or blood-derived products.
5. Any unexpected event relevant to the physician in charge, after discussion with the coordinating investigator and the sponsor

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Change of Transcriptomic profiles | Change from Baseline Transcriptomic profiles at day after vaccine injection (Day 1)
  Transcriptomic profiles of blood cells (microarrays) will be performed to measure early systemic innate immune response
Change of Innate cellular phenotyping | Change from Baseline Innate cellular phenotyping at day after vaccine injection (Day 1)
  Innate cellular phenotyping will be performed using 36 surface markers deciphering lineage cells monocytes, neutrophils, NK, antigen-presenting cells.
Change of Gene signature | Change from Baseline Gene signature at day after vaccine injection (Day 1)
  Study of the transcriptional profile of the blood cells by microarrays
Humoral immune responses | Day 0, Day 21, Day 90 and Day 210 time
  HAI titers, Individual HAI titers ratio, Subjects with titers ≥ 40, Seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: Cecile JANSSEN, Principal Investigator — CH Annecy Genevois
Locations (2):
- France (2):
  - Centre Hospitalier Annecy Genevois, Annecy
  - Centre Hospitalier Métropole Savoie, Chambéry

IPD SHARING:
Plan to Share IPD: No